CLINICAL TRIAL: NCT02611973
Title: French Aspirin Study in Essential Thrombocythemia: an Open and Randomized Study
Brief Title: Hydroxyurea Versus Aspirin and Hydroxyurea in Essential Thrombocythemia
Acronym: FAST
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P140933
Record Dates: First submitted 2015-10-13; First posted 2015-11-23 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: MPN; Essential Thrombocythemia
Keywords: Essential Thrombocythemia; Aspirin
MeSH Terms: conditions — Thrombocythemia, Essential

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HU without aspirin (Experimental)
  Interventions: Other: Aspirin therapy interruption; Drug: Hydroxyurea treatment (HU)
- HU + aspirin maintenance (Active Comparator)
  Interventions: Other: Usual treatment by aspirin 100 mg/d in the active comparator arm; Drug: Hydroxyurea treatment (HU)
- HU + AAG (Other): Observational arm
  Interventions: Other: No interruption of aspirin in the Observational arm; Drug: Hydroxyurea treatment (HU)

INTERVENTIONS:
Other: Aspirin therapy interruption — Stop the treatment by aspirin 100mg/d in the experimental arm.
  Arms: HU without aspirin
Other: Usual treatment by aspirin 100 mg/d in the active comparator arm — HU+ aspirin maintenance
  Arms: HU + aspirin maintenance
Other: No interruption of aspirin in the Observational arm — patient with Contre indication to aspirin or required antithrombotic therapy
  Arms: HU + AAG
Drug: Hydroxyurea treatment (HU) — HU maintenance

SUMMARY:
The hypothesis is that efficient prevention of thrombosis with aspirin at diagnosis becomes less useful once patients have achieved a hematologic response (HR) (modified by amendment 1/03/2017) and/or that this benefit is hampered by an increased hemorrhagic risk especially in elderly patients.

Hence, investigator propose a prospective randomized study to assess the benefit / risk ratio of aspirin maintenance in high risk Essential thrombocythemia (ET) patients, in hematological response (modified by amendment 1/03/2017) on Hydroxyurea.

DETAILED DESCRIPTION:
ET is a myeloproliferative neoplasm (MPN) characterized by a high platelet level. Increased occurrence of thrombosis and hemorrhages are the main complications in ET. In this regard, the key factors defining high risk ET include age over 60 years, past history of thrombosis, platelet > 1500 109/L and to a lesser degree cardiovascular risk factors. These criteria currently serve as therapeutic guidelines for the use of cytoreductive therapy, with hydroxyurea (HU) being the treatment of choice in the first line setting.

The use of antiplatelet agent i.e. low-dose aspirin is also generally recommended. However, the benefit of aspirin has never been formally demonstrated in ET. Only indirect evidence come from the ECLAP study that enrolled patients with polycythemia vera (PV). Of note in the ECLAP study, the efficacy of aspirin was assessed only at diagnosis but not correlated thereafter with the hematological response on cytoreductive therapy.

In general non-MPN population studies, primary prophylaxis with aspirin has been associated with a risk reduction of major vascular events, but an increased risk of hemorrhage, especially considering age and prior gastrointestinal history. In a recent retrospective study, the combination of aspirin and cytoreduction was reported to prevent thrombosis but concomitantly increase the bleeding risk when compared to HU alone , especially in patients older than 60 years, thus questioning the benefits of long term use of aspirin therapy. These data raise the question of the actual benefit of aspirin maintenance, once patients have been efficiently treated with cytoreductive therapy.

Hence, investigator propose a prospective randomized study to assess the benefit / risk ratio of aspirin maintenance in high risk ET patients, in hematological response (modified by amendment 1/03/2017) on Hydroxyurea. Patients for which Aspirin interruption will not be possible because of extra-ET indications will be enrolled in the control observational arm.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years and older (modified by amendment 01/03/2017)
* Contraception considered effective by the investigator: for women of childbearing and for men whose partner is likely to procreate (added by amendment 01/03/2017)

  * Diagnosis of ET performed within the last 10 years (modified by amendment 01/03/2017) : with or without Janus kinase 2V617F (JAK2V617F) mutation according to the WHO 2008 criteria (TEFFERI,2007)
  * ET patients currently treated with hydroxyurea in first line, who have achieved a complete or partial hematologic response according to the ELN 2009 (BAROSI, 2009) modified (at least three month apart and at inclusion) (modified by amendment 01/03/2017)
  * Signed Written Informed Consent
  * Health insurance coverage.

Exclusion Criteria:

* Other myeloproliferative disorder than ET.
* Contra-indication to hydroxyurea.
* Other uncontrolled malignancies at the time of diagnosis or inclusion.
* History of haemostasis perturbation not related to ET, associated with a significant risk of hemorrhage or thrombosis (modified by amendment 01/03/2017)

  -.• Pregnancy or breastfeeding (added by amendment 01/03/2017)
* Inability to freely provide consent through judiciary or administrative condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2250 (Estimated)
Dates: Start 2016-03-10 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of death from vascular origin and other thrombotic and hemorrhagic events (combined endpoint) | at 2-years follow-up
  Definition of vascular events:
  Thrombotic events: Myocardial infarction, unstable angina, stroke, transient ischemic attack, peripheral arterial thrombosis, splanchnic or limb deep vein thrombosis, pulmonary embolism, and erythromelalgia
  Hemorrhagic events:
  Intracranial or retroperitoneal bleed, overt hemorrhage associated with a decrease in hemoglobin ≥20 g/l or overt hemorrhage requiring a blood transfusion of two red blood cell (RBC) units or more, and hemorrhage of grade >=2 according to the NCI Common Toxicity criteria (CTC) V.4.0 scale.
  Deaths will be included as a death from thrombosis or hemorrhage if they satisfied criteria for one of the above diagnoses immediately ANTE-MORTEM or if they had a POST-MORTEM examination confirming the diagnosis. Sudden death of presumed vascular origin without a POST-MORTEM examination will be included as a thrombotic death.

SECONDARY OUTCOMES:
Cumulative incidence and characteristics of vascular complications: thrombosis and hemorrhage, (grade, site, recurrence), assessed yearly over a 5-year follow-up period. | at 5 years
Rate of hematological response every 6 months | at 5 years
  Hematological response as assessed by European Leukemia Net (ELN) criteria, revised ELN International Working Group on Myeloproliferative Neoplasms Research and Treatment (ELN -IWG MRT).
Adverse event (AE) frequency and incidence, comparison in the two arms | at 5 years
Number of HU-related nonhematologic toxicities | at 5 years
Cumulative incidence of thrombosis | at 5 years
Cumulative incidence of hemorrhagic complications | at 5 years
Estimation of the progression-free survival | at 5 years
Estimation of overall survival | at 5 years
Short Form 36 (SF36) Health Survey | through study completion, an average of 1 year
  Evaluation of quality of life by using SF36
Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) | through study completion, an average of 1 year
  Evaluation of quality of life by using (MPN-SAF)
Number of mortality cause. | at 5 years
Cumulative incidence of progression to polyglobulia | at 5 years
Cumulative incidence of progression to myelofibrosis (MF) | at 5 years
Cumulative incidence of progression to myelodysplastic syndrome (MDS) | at 5 years
Cumulative incidence of progression AML | at 5 years
Frequencies of mutations (JAK2V617F, MPLw515 and CALR) and JAK2V617F allele burden, MPLw515 allele burden and CALR mutation allele burden (in blood DNA) in patients presenting thrombosis or not . | at 5 years
Frequencies of mutations (JAK2V617F, MPLw515 and CALR) and JAK2V617F allele burden, MPLw515 allele burden and CALR mutation allele burden in patients in persistent hematological response (modified by amendment 1/03/2017). | at 5 years
  responses and intolerance define according to ELN criteria
Frequencies of mutations (JAK2V617F, MPLw515 and CALR) and JAK2V617F allele burden, MPLw515 allele burden and CALR mutation allele burden in patient who will lose their hematological response (modified by amendment 1/03/2017). | at 5 years
  responses and intolerance define according to ELN criteria
Frequencies of mutations (JAK2V617F, MPLw515 and CALR) and JAK2V617F allele burden, MPLw515 allele burden and CALR mutation allele burden in patients presenting intolerance to treatment. | at 5 years
  responses and intolerance define according to ELN criteria

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Giraudier, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Background] Alvarez-Larran A, Pereira A, Arellano-Rodrigo E, Hernandez-Boluda JC, Cervantes F, Besses C. Cytoreduction plus low-dose aspirin versus cytoreduction alone as primary prophylaxis of thrombosis in patients with high-risk essential thrombocythaemia: an observational study. Br J Haematol. 2013 Jun;161(6):865-71. doi: 10.1111/bjh.12321. Epub 2013 Apr 12. PMID 23577924
- [Background] Barbui T, Barosi G, Birgegard G, Cervantes F, Finazzi G, Griesshammer M, Harrison C, Hasselbalch HC, Hehlmann R, Hoffman R, Kiladjian JJ, Kroger N, Mesa R, McMullin MF, Pardanani A, Passamonti F, Vannucchi AM, Reiter A, Silver RT, Verstovsek S, Tefferi A; European LeukemiaNet. Philadelphia-negative classical myeloproliferative neoplasms: critical concepts and management recommendations from European LeukemiaNet. J Clin Oncol. 2011 Feb 20;29(6):761-70. doi: 10.1200/JCO.2010.31.8436. Epub 2011 Jan 4. PMID 21205761
- [Background] Barosi G, Birgegard G, Finazzi G, Griesshammer M, Harrison C, Hasselbalch HC, Kiladjian JJ, Lengfelder E, McMullin MF, Passamonti F, Reilly JT, Vannucchi AM, Barbui T. Response criteria for essential thrombocythemia and polycythemia vera: result of a European LeukemiaNet consensus conference. Blood. 2009 May 14;113(20):4829-33. doi: 10.1182/blood-2008-09-176818. Epub 2009 Mar 10. PMID 19278953
- [Background] Barosi G, Mesa R, Finazzi G, Harrison C, Kiladjian JJ, Lengfelder E, McMullin MF, Passamonti F, Vannucchi AM, Besses C, Gisslinger H, Samuelsson J, Verstovsek S, Hoffman R, Pardanani A, Cervantes F, Tefferi A, Barbui T. Revised response criteria for polycythemia vera and essential thrombocythemia: an ELN and IWG-MRT consensus project. Blood. 2013 Jun 6;121(23):4778-81. doi: 10.1182/blood-2013-01-478891. Epub 2013 Apr 16. PMID 23591792
- [Background] Barosi G, Birgegard G, Finazzi G, Griesshammer M, Harrison C, Hasselbalch H, Kiladijan JJ, Lengfelder E, Mesa R, Mc Mullin MF, Passamonti F, Reilly JT, Vannucchi AM, Barbui T. A unified definition of clinical resistance and intolerance to hydroxycarbamide in polycythaemia vera and primary myelofibrosis: results of a European LeukemiaNet (ELN) consensus process. Br J Haematol. 2010 Mar;148(6):961-3. doi: 10.1111/j.1365-2141.2009.08019.x. Epub 2009 Nov 23. No abstract available. PMID 19930182